CLINICAL TRIAL: NCT02671552
Title: Contrast-Enhanced Ultrasound for the Evaluation of Renal Cell Carcinoma Cryoablation
Brief Title: Contrast-Enhanced Ultrasound in Predicting Treatment Response in Patients With Kidney Cancer Undergoing Cryosurgery
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Terminated by the IRB
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12P.615; 2012-84 (Other: Thomas Jefferson University); NCI-2015-01470 (Registry Identifier: NCI Clinical Trials Reporting Program); JT 3004 (Other: JeffTrial Number)
Record Dates: First submitted 2016-01-04; First posted 2016-02-02 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diagnostic (contrast-enhanced ultrasound) (Experimental): Patients receive perflutren protein-type A microspheres IV and then undergo contrast-enhanced ultrasound imaging the morning prior to cryosurgery and at 3-4 months post treatment during Magnetic Resonance Imaging (MRI) or computed tomography (CT) follow up.
  Interventions: Drug: Perflutren Protein-Type A Microspheres; Procedure: Dynamic Contrast-Enhanced Ultrasound Imaging

INTERVENTIONS:
Drug: Perflutren Protein-Type A Microspheres — Given IV
  Other Names: Optison, Perflutren Protein-Type A Microspheres
Procedure: Dynamic Contrast-Enhanced Ultrasound Imaging — Undergo contrast-enhanced ultrasound imaging

SUMMARY:
This pilot clinical trial compares the imaging results of contrast-enhanced ultrasound to contrast-enhanced magnetic resonance imaging (MRI) or computed tomography (CT), the current clinical standard, in predicting treatment response in patients with kidney cancer undergoing cryosurgery (a procedure in which an extremely cold liquid or an instrument called a cryoprobe is used to freeze and destroy abnormal tissue). Using contrast-enhanced ultrasound that does not involve a dye may help patients avoid side effects from a dye that is usually used in MRI or CT and may help doctors measure blood flow and determine whether the cryosurgery procedure treated the kidney tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate if contrast-enhanced ultrasound can be used to successfully evaluate the cryoablation (cryosurgery) of renal cell carcinoma.

SECONDARY OBJECTIVES:

I. Establish whether contrast-enhanced ultrasound provides a reliable tool for the characterization of renal masses prior to cryoablation.

TERTIARY OBJECTIVES:

I. Compare harmonic imaging (the current industry standard for contrast imaging) with subharmonic imaging (a novel, improved contrast imaging technique) in the two aims listed above.

OUTLINE:

Patients receive perflutren protein-type A microspheres intravenously (IV) and then undergo contrast-enhanced ultrasound imaging the morning prior to cryosurgery and at 3-4 months post treatment during MRI or CT follow up.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for a percutaneous cryoablation of a renal mass
* Be medically stable
* If a female of child-bearing potential, must have a negative pregnancy test
* Have signed informed consent to participate in the study

Exclusion Criteria:

* Females who are pregnant or nursing
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable; for example:

  * Patients on life support or in a critical care unit
  * Patients with unstable occlusive disease (eg, crescendo angina)
  * Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia
  * Patients with uncontrolled congestive heart failure (New York Heart Association [NYHA] class IV)
* Patients with recent cerebral hemorrhage
* Patients with known sensitivities to albumin, blood, or blood products
* Patients who have undergone surgery within 24 hours prior to the study sonographic examination
* Patients with known hypersensitivity to perflutren
* Patients who have received any contrast medium (X-ray, MRI, CT, or ultrasound [US]) in the 24 hours prior to the research US exam
* Patients with cardiac shunts
* Patients with congenital heart defects
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli
* Patients with respiratory distress syndrome
* Patients with renal insufficiency such that they can not get intravenous contrast as part of screening or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2014-12-04 (Actual); Study Completion 2014-12-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Sensitivity will be calculated for the contrast-enhanced ultrasound exam using both the standard of care contrast-enhanced CT or MRI, and patient outcome as the reference standard. Correlations between these findings and both contrast-enhanced MRI or CT findings and patient outcomes will be compared using the Fisher exact test.
Specificity - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Specificity will be calculated for the contrast-enhanced ultrasound exam using both the standard of care contrast-enhanced CT or MRI, and patient outcome as the reference standard. Correlations between these findings and both contrast-enhanced MRI or CT findings and patient outcomes will be compared using the Fisher exact test.
Accuracy - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Accuracy will be calculated for the contrast-enhanced ultrasound exam using both the standard of care contrast-enhanced CT or MRI, and patient outcome as the reference standard. Correlations between these findings and both contrast-enhanced MRI or CT findings and patient outcomes will be compared using the Fisher exact test.
Positive predictive value - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Positive predictive value will be calculated for the contrast-enhanced ultrasound exam using both the standard of care contrast-enhanced CT or MRI, and patient outcome as the reference standard. Correlations between these findings and both contrast-enhanced MRI or CT findings and patient outcomes will be compared using the Fisher exact test.
Negative predictive value - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Negative predictive value will be calculated for the contrast-enhanced ultrasound exam using both the standard of care contrast-enhanced CT or MRI, and patient outcome as the reference standard. Correlations between these findings and both contrast-enhanced MRI or CT findings and patient outcomes will be compared using the Fisher exact test.

SECONDARY OUTCOMES:
Sensitivity - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Inter- and intra-observer variability will be calculated.
Specificity - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Inter- and intra-observer variability will be calculated.
Positive predictive value - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Inter- and intra-observer variability will be calculated.
Negative predictive value - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Inter- and intra-observer variability will be calculated.
Accuracy - Ability of contrast-enhanced ultrasound to successfully evaluate the cryoablation of renal cell carcinoma | Up to 3-4 months after cryosurgery
  Inter- and intra-observer variability will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/